CLINICAL TRIAL: NCT01024998
Title: A Phase 1, Open-Label, Multi-Center, Dose-Escalating, Safety and Tolerability Study of a Single Intravitreal Injection of AAV2-sFLT01 in Patients With Neovascular Age-Related Macular Degeneration
Brief Title: Safety and Tolerability Study of AAV2-sFLT01 in Patients With Neovascular Age-Related Macular Degeneration (AMD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: sFLT01-AMD-00106; 0810-948 (Other: NIH Office of Biotechnology Activities); MSC12870 (Other: Sanofi)
Record Dates: First submitted 2009-12-02; First posted 2009-12-03 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Macular Degeneration; Age-Related Maculopathies; Age-Related Maculopathy; Maculopathies, Age-Related; Maculopathy, Age-Related; Retinal Degeneration; Retinal Neovascularization; Gene Therapy; Therapy, Gene; Eye Diseases
Keywords: Age-Related Macular Degeneration; AMD; Wet AMD; Neovascular AMD; Ocular; Ocular gene therapy; Subretinal neovascularization
MeSH Terms: conditions — Macular Degeneration; Retinal Degeneration; Retinal Neovascularization; Eye Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 2 x 10^8 vector genomes (vg) AAV2-sFLT01 (Experimental)
  Interventions: Biological: AAV2-sFLT01
- 2 x 10^9 vector genomes (vg) AAV2-sFLT01 (Experimental)
  Interventions: Biological: AAV2-sFLT01
- 6 x 10^9 vector genomes (vg) AAV2-sFLT01 (Experimental)
  Interventions: Biological: AAV2-sFLT01
- 2 x 10^10 vector genomes (vg) AAV2-sFLT01 (Experimental)
  Interventions: Biological: AAV2-sFLT01

INTERVENTIONS:
Biological: AAV2-sFLT01 — 2 x 10^8 vector genomes (vg) AAV2-sFLT01. Single intravitreal injection to a single eye, using a fixed volume of 100 μL.
  Arms: 2 x 10^8 vector genomes (vg) AAV2-sFLT01
Biological: AAV2-sFLT01 — 2 x 10^9 vector genomes (vg) AAV2-sFLT01. Single intravitreal injection to a single eye, using a fixed volume of 100 μL.
  Arms: 2 x 10^9 vector genomes (vg) AAV2-sFLT01
Biological: AAV2-sFLT01 — 6 x 10^9 vector genomes (vg) AAV2-sFLT01. Single intravitreal injection to a single eye, using a fixed volume of 100 μL.
  Arms: 6 x 10^9 vector genomes (vg) AAV2-sFLT01
Biological: AAV2-sFLT01 — 2 x 10^10 vector genomes (vg) AAV2-sFLT01. Single intravitreal injection to a single eye, using a fixed volume of 100 μL.
  Arms: 2 x 10^10 vector genomes (vg) AAV2-sFLT01

SUMMARY:
This Phase 1 clinical research study will examine the safety and tolerability of an experimental gene transfer agent, AAV2-sFLT01, in patients with Neovascular Age-Related Macular Degeneration (AMD).

DETAILED DESCRIPTION:
A new treatment for neovascular age-related macular degeneration (AMD) is being investigated. Neovascular AMD is sometimes referred to as the "wet" form of AMD. The purpose of this Phase 1 clinical research study is to examine the safety and ability of an experimental study drug to treat a complication of the disease which leads to vision loss. The name of the study drug is "AAV2-sFLT01." This experimental study drug uses a virus to transfer a gene (genetic code) into cells within the eye. The gene codes for a protein that is intended to diminish the growth of abnormal blood vessels under the retina. The duration of the gene's effect is currently unknown, but might last for years.

This clinical research study will look at the safety of a single administration of AAV2-sFLT01 injected directly into the eye. There are 2 parts to this study, but patients will take part in only one of them. In the first part of the study, 4 different doses of the study drug will be studied in 4 separate groups of patients. Patients in the first part of the study will not be randomized. In the second part of the study, the highest dose that was safe and well tolerated will be studied in 10 more patients. Patients in this part of the study may have a ranibizumab (Lucentis®) injection 26 weeks after their AAV2-sFLT01 injection to verify their responsiveness to anti-VEGF therapy, if they have not demonstrated a response to AAV2-sFLT01. The initial two parts of this protocol are expected to be completed in July, 2013.

All patients injected with AAV2-sFLT01 will be asked to participate in an Extended Follow-Up (EFU) program for up to an additional 4 years. Participation is voluntary but strongly encouraged as it allows for the long term collection of safety information as well as information about the potential long term effects of the study drug. Study visits will take place at the site every 6 months.

Up to thirty-four (34) patients at multiple centers will take part in this study in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Choroidal neovascular membrane (CNV) secondary to AMD, as confirmed by the patient's medical history and a documented diagnosis of CNV.
* Distance BCVA of 20/100 or worse in the study eye.
* The fellow eye must have distance BCVA of 20/400 or better.
* The study eye, i.e., the eye that receives investigational product, has the worst CVA (As compared to the fellow eye).
* Subfoveal disciform scarring in the study eye for the first part of the study (the dose-escalation part). Patients may or may not have macular scarring in the study eye for the second part of the study (MTD phase). In addition, patients enrolled in the second part of the study must have demonstrated responsiveness to an anti-VEGF therapy within 12 months prior to screening and after the patient's most recent treatment of anti-VEGF therapy.
* Noted presence of intra- or sub-retinal fluid.
* Adequate dilation of pupils to permit thorough ocular examination and testing.
* Must be willing to have samples of anterior chamber fluid collected from the study eye.

Exclusion Criteria:

* CNV in the study eye due to any reason other than AMD.
* History of conditions in the study eye during Screening which might alter visual acuity or interfere with study testing.
* Active uncontrolled glaucoma.
* Had any intraocular surgeries in the study eye within 3 months of enrollment or are known or likely candidates for intraocular surgery (including cataract surgery) in the study eye within 1 year of treatment.
* Acute or chronic infection in the study eye.
* History of inflammation in the study eye or ongoing inflammation in either eye.
* Any contraindication to intravitreal injection.
* Received Photo Dynamic Therapy in the study eye within 60 days, or laser photocoagulation within 14 days prior to Screening.
* Currently using or have used ranibizumab (Lucentis®), bevacizumab (Avastin™), or pegaptanib sodium (Macugen®) within 1 month prior to Screening.
* Currently using or have used Aflibercept (Eylea®) within 4 months prior to Screening.
* Currently using any periocular (study eye), intravitreal (study eye), or systemic (oral or intravenous) steroids within 3 months prior to Screening.
* Any active herpetic infection, in particular active lesions in the eye or on the face.
* Any significant poorly controlled illness that would preclude study compliance and follow-up.
* Current or prior use of any medication known to be toxic to the retina or optic nerve.
* Previous treatment with any ocular or systemic gene transfer product.
* Received any investigational product within 120 days prior to Screening.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-01-11 (Actual); Primary Completion 2014-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of a single uniocular intravitreal injection of AAV2-sFLT01 | Time of treatment through Week 52 (referred to as the "core" study)
Number of Treatment Emergent Adverse Events | Time of treatment through Week 52 (referred to as the "core" study)
Number of Treatment Emergent Adverse Events | Up to 4 years after the "core" study (referred to as the "Extended Follow-up" period)

SECONDARY OUTCOMES:
Decreased retinal thickness | Time of treatment through Week 52 (referred to as the "core" study)
Decreased retinal thickness | Up to 4 years after the "core" study (referred to as the "Extended Follow-up" period)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (4):
- United States (4):
  - investigational site number 03WilmerEy, Baltimore, Maryland
  - investigational site number 02Ophthalm, Boston, Massachusetts
  - investigational site number 01UMassMem, Worcester, Massachusetts
  - investigational site number 05RetinaCo, Slingerlands, New York

REFERENCES:
- [Derived] Heier JS, Kherani S, Desai S, Dugel P, Kaushal S, Cheng SH, Delacono C, Purvis A, Richards S, Le-Halpere A, Connelly J, Wadsworth SC, Varona R, Buggage R, Scaria A, Campochiaro PA. Intravitreous injection of AAV2-sFLT01 in patients with advanced neovascular age-related macular degeneration: a phase 1, open-label trial. Lancet. 2017 Jul 1;390(10089):50-61. doi: 10.1016/S0140-6736(17)30979-0. Epub 2017 May 17. PMID 28526489